CLINICAL TRIAL: NCT04992416
Title: Immediately Placed Implants Using Simvastatin and Autogenous Tooth Graft Combination in Periodontally Compromised Sites: A Randomized Controlled Clinical Trial
Brief Title: Immediately Placed Implants Using Simvastatin and Autogenous Tooth Graft Combination in Periodontally Compromised Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, Principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-27
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Autogenous Tooth Bone Graft; Immediate Implant Placement; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMV with ATBG around implant (Experimental): SMV mixed with ATBG around immediately placed dental implants in the extraction sockets
  Interventions: Procedure: immediate implant placement with ATBG and SMV
- ATBG around implant (Active Comparator): ATBG around immediately placed dental implants in the extraction sockets
  Interventions: Procedure: immediate implant placement with ATBG

INTERVENTIONS:
Procedure: immediate implant placement with ATBG and SMV — immediate implant placement using ATBG as a graft material, with SMV
  Arms: SMV with ATBG around implant
Procedure: immediate implant placement with ATBG — immediate implant placement using ATBG as a graft material without SMV
  Arms: ATBG around implant

SUMMARY:
Recently, autogenous tooth graft (ATG) made from compromised teeth was applied in bone defects and resulted in a good clinical efficacy.(6) Moreover, it is more accepted by patients to use extracted teeth as a bone graft material, especially in the case of immediate implant placement. Simvastatin (SMV), known as a 3-hydroxy-3-methylglutaryl-CoA (HMG-CoA) reductase inhibitor, is widely used to decrease serum cholesterol because of its safe and effective treatment. Apart from cholesterol-lowering effects, SMV is also found to promote osteogenic differentiation of bone marrow stem cells (BMSCs), suppress osteoclastic differentiation in bone tissue and promotes osseointegration around implants in animal studies. SMV is reported to enhance autophagy and alleviates the ROS of BMSCs in the osseointegration of implants. The present study will be carried out to evaluate the effect of SMV combined with ATG on bone formation around immediately placed dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Teeth need to be extracted for periodontal reasons with a defect of labial bone (horizontal or vertical bone defect).
* the teeth without acute inflammation.
* no uncontrolled systemic disease which is not suitable for implantation.
* Good systemic and oral health.

Exclusion Criteria:

* patients with systemic diseases or medications known to alter healing processes.
* Psychiatric disorders.
* Root canal treated teeth.
* patients undergoing or who had undergone radiation therapy and chemotherapy to the head and neck region during 12 months.
* patients with para-functional habits.
* alcoholics.
* drug abusers.
* heavy smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
clinical evaluation of bone formation around immediately placed dental implants | 9 months
  Changes on bone formation using ATBG with or without SMV around immediately placed dental implants in periodontally compromised teeth
radiographic outcome around immediately placed dental implants | 9 months
  the radiographic outcome of ATBG on bone formation with or without SMV around immediately placed dental implants in periodontally compromised teeth

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt

REFERENCES:
- [Derived] Issa DR, Nassar M, Elamrousy W. Immediately placed implants using simvastatin and autogenous tooth graft combination in periodontally compromised sites: a randomized controlled clinical trial. Clin Oral Investig. 2024 Mar 12;28(4):210. doi: 10.1007/s00784-024-05596-4. PMID 38467945